CLINICAL TRIAL: NCT03058614
Title: Contrast-enhanced Ultrasound Versus CT Scan for Kidney Stone Patient
Brief Title: Contrast-enhanced Ultrasound Versus CT Scan for Kidney Stone Patient Management
Acronym: CEUS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The research team submitted grants over the course of several years to gain funds to support this research but were unsuccessful in securing the funds. The research team will now focus on other funded studies.
Sponsor: University of California, San Francisco (Other)
Collaborators: Oregon Health and Science University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Thomas Chi, MD, Assistant Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 17-21497; R21DK109433 (NIH)
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Ultrasonography; Nephrolithiasis
Keywords: Contrast-enhanced ultrasound; Percutaneous nephrolithotomy
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Intervention Model Description: Randomized control study
Who Masked: Care Provider, Investigator
Masking Description: The surgical team will be blinded to the randomization outcome of the patient until the day after surgery so as to minimize any bias introduced into their preoperative counseling. After that point, treatment teams will no longer be blinded to randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CEUS arm (Active Comparator): On postoperative day 1 (unless not clinically indicated), each subject will undergo CEUS with an administration of Lumason via their pre-placed nephrostomy tube.
  Interventions: Drug: CEUS
- CT scan plus capping trial arm (Active Comparator): On postoperative day 1 (unless not clinically indicated), subjects' pre-placed nephrostomy tube will be capped and they will undergo a low dose non-contrast abdominal CT scan.
  Interventions: Diagnostic Test: Non-contrast CT scan; Diagnostic Test: Capping trial

INTERVENTIONS:
Drug: CEUS — In subjects randomized into the CEUS arm, 2 mL of Lumason will be injected as a single dose via a nephrostomy tube at the time of postoperative renal ultrasound, following by 5 mL of normal saline flush. Subjects will be given up to one additional dose injected in the same fashion as indicated during the imaging study to confirm opacification of the ureter.
  Other Names: Contrast-enhanced ultrasound, CEUS nephrostogram
  Arms: CEUS arm
Diagnostic Test: Non-contrast CT scan — The CT scan performed in this study arm is regularly performed to evaluate the kidney and look for residual stones after surgery both at UCSF and around the world. It does not require contrast injection, so risks from contrast allergy or any injection are absent. A low dose protocol will be used, and therefore, subjects will be exposed to a very small amount of ionizing radiation as low as 1-2 mSv if randomized into this arm.
  Other Names: NCCT
  Arms: CT scan plus capping trial arm
Diagnostic Test: Capping trial — Subjects who are randomized into this study arm will undergo both nephrostomy tube capping and a low dose non-contrast CT scan on the first day after surgery. Successfully passing a capping trial is defined as the absence of fever, worsened flank pain, and leakage around the nephrostomy tube within 4 hours after capping the tube.
  Arms: CT scan plus capping trial arm

SUMMARY:
This study will be a randomized controlled study comparing the use of two clinical management strategies in nephrostomy tube management following percutaneous nephrolithotomy (PCNL). The first strategy entails using contrast-enhanced ultrasound (CEUS) to evaluate the renal collecting system (1). This is a new imaging approach applying ultrasound machines with special software in combination with intraluminal ultrasound contrast agent (Lumason) injection, which is an FDA-approved ultrasound contrast agent (2). The second strategy is a nephrostomy tube capping trial combined with low dose non-contrast computed tomography (CT) scan, one of the most frequently utilized clinical management strategies currently used in clinical practice (3).

DETAILED DESCRIPTION:
This is a multi-center, randomized controlled study comparing the use of CEUS to CT scan plus capping trial immediately following PCNL. A total recruitment target of 1,046 subjects is planned and participants will be randomized into one of the two study arms.

1. Contrast-enhanced ultrasound (CEUS) arm: On postoperative day 1 (unless not clinically indicated), each subject will undergo CEUS with an administration of Lumason via their pre-placed nephrostomy tube.
2. Non-contrast CT scan plus capping trial arm: On postoperative day 1 (unless not clinically indicated), subjects' pre-placed nephrostomy tube will be capped and they will undergo a low dose non-contrast abdominal CT scan.

Subsequently, nephrostomy tubes will be managed based on the results from these studies by the treating surgeon.

Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study.

The following investigational regimen will be used only in the CEUS arm:

Experimental Investigation: Lumason at a 2 mL single dose, repeatable once at the time of imaging as needed.

Subjects will be exposed to the randomization schema for 1 day during which they will undergo one of the two diagnostic imaging pathways. After that imaging study is complete, clinical care will proceed as per norm. Clinical and imaging data will be prospectively collected from the time of initial presentation until 6 months after surgery. The total duration of the study is expected to be 5 years to reach target accrual. Therefore, the investigators anticipate that the total duration of this study will be 4 years and 6 months for patient recruitment with the final 6 months used for collecting follow up data.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older.
* Renal and/or ureteral stone of any size diagnosed either by ultrasound or CT scan and requiring surgical treatment with percutaneous removal (PCNL).

Exclusion Criteria:

* A second stage PCNL is planned or expected after surgery, entailing that postoperative tube management is pre-determined.
* Subjects with serious illness likely to cause death within the next 5 years, so as to exclude significant metabolic derangements that might lead to adverse surgical outcome.
* Subjects with a history of hypersensitivity reactions to sulfur hexafluoride lipid microsphere components or to any of the inactive ingredients in Lumason
* Pregnancy, which is a contraindication to both CT scan and ultrasound contrast injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-30 (Estimated); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Radiation exposure dose | 6 months following surgery
  For radiation exposure dose measurement in this study, the investigators will use dose metrics obtained from the Digital Imaging and Communications within the scanners or Picture Arching and Communication system (PACS).

SECONDARY OUTCOMES:
Rate of adverse clinical events | 6 months following surgery
  Defined as postoperative complications and any unplanned surgery related to the patient's kidney stone

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Chi, MD, Principal Investigator — UCSF Department of Urology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chi T, Usawachintachit M, Mongan J, Kohi MP, Taylor A, Jha P, Chang HC, Stoller M, Goldstein R, Weinstein S. Feasibility of Antegrade Contrast-enhanced US Nephrostograms to Evaluate Ureteral Patency. Radiology. 2017 Apr;283(1):273-279. doi: 10.1148/radiol.2016160959. Epub 2016 Oct 19. PMID 28234551
- [Background] Lumason: Prescribing Information [Internet]. [cited 2017 Jan 21]. Available from: http://www.braccoimaging.com/us-en/products-and-solutions/contrast-enhanced-ultrasound/lumason/prescribing-information
- [Background] Sountoulides P, Metaxa L, Cindolo L. Is computed tomography mandatory for the detection of residual stone fragments after percutaneous nephrolithotomy? J Endourol. 2013 Nov;27(11):1341-8. doi: 10.1089/end.2012.0253. Epub 2013 Jul 9. PMID 23590513